CLINICAL TRIAL: NCT04073862
Title: Assessing Feasibility of Stepped Care TF-CBT in Norwegian Municipalities
Brief Title: The Norwegian Stepped-Care TF-CBT Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-TF-CBT-pilot
Record Dates: First submitted 2019-06-03; First posted 2019-08-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Post Traumatic Stress Disorder (PTSD); Depressive Symptoms; Parental Stress; Health Related Quality of Life
Keywords: Stepped-Care Trauma-Focused Cognitive Behavioral Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Intervention Model Description: Upon training in SC-TF-CBT, therapists in Norwegian municiplaities across the country will administer the treatment as deemed appropriate. Data will be collected to determine feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stepped-Care TF-CBT (Other): The study participants will receive Stepped-Care Trauma-Focused Cognitive-Behavioral-Therapy (SC-TF-CBT).
  Interventions: Other: Stepped-Care TF-CBT

INTERVENTIONS:
Other: Stepped-Care TF-CBT — SC-TF-CBT will be administered to children meeting the inclusion criteria of the study. The treatment aims to improve daily function for trauma-exposed children and their families by way of stress-mastery exercises, coping skills and gradual exposure.

SUMMARY:
Every day, a significant number of children and young people in Norway experience violence, abuse, or other potentially traumatizing events. These children are at risk of developing serious health problems such as post-traumatic stress disorder (PTSD), anxiety, depression, behavioral problems, and drug dependency. Moreover, when left unaddressed, trauma experiences in childhood can have long-term implications for work- and educational participation as well as later subjection to violence. Provision of accessible and situationally adaptable treatments can therefore have great benefits for children, families, and communities at large.

In this project, the investigators will introduce the method of Stepped-Care Trauma-Focused Behavioral Cognitive Therapy (SC-TF-CBT) in a selection of 15 municipalities across Norway. SC-TF-CBT is a parent-led - therapist-assisted low-threshold method aimed at treating children exposed to abuse, sexual assault, or other trauma and who are at risk of developing more severe trauma-related difficulties (Salloum, et al. 2014). This is the first test of the method outside the US. The project's main aim is therefore to evaluate the feasibility and efficiency of the treatment in a Norwegian context through a pre-post design.

The following questions are to be explored:

1. How does the SC-TF-CBT model fit the Norwegian health care culture and service system?
2. When testing Stepped-Care in a Norwegian context, the model is set to involve both the municipal and specialist service levels. Severe cases will be stepped up/transferred to the specialist level for TF-CBT treatment. How do these transitions work for the participating families, and what are the experiences and perspectives of practitioners and service-leaders regarding coordination and collaboration between service levels?
3. Do the children, parents, and therapists like working with the method?
4. Do recipients of the treatment (children and parents) report symptom improvement?
5. Which children and parents seem to benefit the most from the method, and who do not?

DETAILED DESCRIPTION:
Stepped-Care Trauma-Focused Behavioral Cognitive Therapy (SC-TF-CBT) is a semi home-based treatment for children at risk of developing PTSD, where the child's caregiver takes on the role as helper under the guidance of a trained therapist. The treatment runs over a course of approximately 12-15 weeks and has two phases. In cases where symptom improvement is evident after 6-9 weeks, the following 6 weeks is a maintenance phase. In the maintenance phase, the child and caregiver will continue with some of the exercises found helpful and engage in pleasant activities together, while receiving follow-ups by the therapist.

In cases where symptoms persist, however, the treatment is stepped up to TF-CBT. In the Norwegian context, in contrast to the US, stepping up will imply that responsibility for the treatment is transferred from the municipal service level to a Child and Youth Psychiatric Policlinic (BUP). In this particular way, the treatment scheme is adapted to the local context, while ensuring continuity as intended by the developers. Examining how this transition is experienced, how the transition is reasoned for and organized, and the transitions correspond with treatment needs are therefore important objectives.

The first stage of this trial project involves providing SC-TF-CBT training to 45 therapists (primarily clinical psychologists with experience in trauma treatment and working with children/ families) in the 15 municipalities across Norway. Training is carried out by specialists in psychology at NKVTS in collaboration with the University of South Florida (USF). Following the training, the therapists will receive referrals as usual, but will be equipped with an additional treatment method.

While protocols exist for two age categories (3-6 and 7-12), this project focuses on children between the ages of 7-12. In total, about 80 children (and caregivers) will participate in the study. This estimate takes into account a possible dropout rate of about 30 percent. In order to produce sufficiently strong analysis, including mediator analyses, the investigators' calculations indicate that the study requires 58 children to complete the SC-TF-CBT program. Based on current data and rate of missingness, the earlier estimate of 75 participants has been changed to 80 (Nov.2021).

Caregivers and children participating in the study will be asked to provide information about symptoms and treatment experiences at several points throughout the treatment trajectory. The therapist will collect information by way of assessment forms available for completion on iPads. The therapists will also submit evaluations throughout the trajectory of each family by way of online assessment forms and 3 months after treatment completion. Audio recordings from treatment session will be used to determine fidelity.

To attain data on entire trajectories, from pre-screening through completed treatments, the quantitative data will be supplemented by qualitative, semi-structured interviews with children, caregivers, and therapists. The interviews are to take place upon treatment completion, after approximately 12-15 weeks. A similar time-frame will be adopted for interviews with families transferred to the specialist service level, who will complete one interview after completion/interruption of Step 1, and then a short second interview 12 weeks after starting treatment in specialist health services, to explore the experiences with the transition. Additionally, to assess the long-term effects of the treatment, the investigators will invite a sample of children and caregivers for follow-up interviews 3-4 months after completion.

Hypotheses:

For research questions 1-3 we expect that most children, caregivers, therapists, and municipality leaders will find the model suitable and acceptable, however, we also expect that some aspects will be perceived as challenging, and that there may be need for adjustments in both the material and strategy for implementation.

For research question 4, it is hypothesized that:

* Children will report lower symptom levels (PTSS, depressive symptoms) and better functioning and quality of life (CGI, 17D) after the completion of step one.
* Parents will report lower symptom levels (PTSS, anxiety, depression), reduced parental stress, and increase in positive aspects of being a parent after the completion of step one.

For research question 5 it is hypothesized that:

* Children exposed to several traumatic events will be at higher risk of non-response compared to children exposed to fewer traumatic events.
* Children exposed to interpersonal trauma will be at higher risk of non-response compared to children exposed to non-interpersonal trauma.
* Higher levels of child PTSS, depression, and posttraumatic cognitions pre-treatment predicts non-response.
* Higher levels of parents' PTSS, anxiety, depression, and negative emotional reactions related to the child's trauma pre-treatment will predict dropout and non-response.
* Lower levels of parents' perceived social support and less percceived positive aspects of being a parent pre-treatment will predict dropout and non-response.
* More barriers and lower expectations to the treatment by parents will predict dropout and non-response.
* Changes in parents' mental health (PTSS, anxiety, depression), emotional reactions and perceived positive aspects of being a parent will predict subsequent change in the child's general functioning, depressive symptoms, and quality of life, but will not predict changes in child's level of PTSS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-12
2. Exposure to at least one episode of violence or other potentially traumatizing event
3. At least 3 years old at time of trauma
4. Minimum 5 symptoms of PTSS (i.e., a frequency score of 2 or 3 on the CATS) of which at least 1 symptom is reexperiencing and 1 symptom is avoidance
5. The therapist must talk to the child alone to make sure that the child is safe at home (see exclusion criteria)
6. At least one month has passed since the last traumatic event.

In addition:

A. If two or more siblings fulfill the inclusion criteria, only the youngest should be included in the study

Exclusion Criteria:

1. Suspicions of psychosis, mental retardation, autism spectrum disorder in the child or any condition that would limit the caregiver's ability to understand CBT and the child's ability to follow instructions.
2. Not fluent in Norwegian and needs interpreter to complete treatment
3. The caregiver who would be treatment participant was the perpetrator, or perpetrator still living at home
4. Parent has had substance use disorder (SUD) within the past 3 months.
5. Child or caregiver is suicidal
6. If child is taking psychotropic medication regimen must be stable for 4 weeks. However, for stimulants or benzodiazepines, the medication regimen must be stable for 2 weeks.
7. Child is currently receiving an other type of trauma treatment

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
CATS 2.0 (Children version / Caregiver version) - Assessment of Change in Symptoms | Baseline (T0), 6-9 weeks (T2), 12-15 weeks (T3), 24-27 weeks (T4)
  Clinical Assessment of Trauma Paths and Symptoms (CATS) (Sachser et al., 2017). The investigators use a revised edition of CATS, based on DSM5 and ICD-11. CATS consists of 15 questions about stressful or scary experiences, 20 questions measuring level of post-traumatic stress responses (to be answered if "yes" on one of the first 15 items), and 5 questions about the social/ performance consequences of experienced problems. Both the Children's version and the Caregiver version of CATS 2.0 contain the same questions, but formulated according to their different points of view. The 15 questions about trauma events are answered by indicating "yes" or "no." The 20 items about symptomatology are scored from 0 (never) to 3 (almost all the time). The final 5 items are indicated with "yes" or "no." In order to measure change, the questions will be completed at three points in time by caregivers and children, respectively.

SECONDARY OUTCOMES:
Quality of life in pre-adolescence: a 17-dimensional health-related measure (17D) | T1 (start-up), 6-9 weeks (T2), T3 (12-15 weeks), 24-27 weeks (T4)
  17D is a validated health-related quality of life survey for children aged 8-11 years (but can be used for 7-year-olds with the aid of an adult) (Apajasalo et al., 1996). The form consists of 17 questions that deal with both physical and mental health. On each of the 17 questions (dimensions) the respondent indicates the appropriate level on each dimension). The scale runs from 1-5, with 5 indicating better outcome. Each dimension has been ascribed a utility weight, which is used to calculate an overall score across dimensions. Quality of life is determined by a single index (17D score) on a 0-1 scale, where 1 is the better outcome.
Acceptability of Intervention Measure (AIM) | Baseline (T0)
  Acceptability of Intervention Measure (AIM) is one of three related instruments (acceptability, appropriateness, and feasibility) developed to fill a need for measures to predicting outcomes, for instance when a treatment is about to be introduced in a new context (Weiner et al., 2017). According to the developers, the measures can be used together or separately. The present research will use the measures, which are scored separately, together to predict how Stepped-Care TF-CBT might suit a Norwegian context. Translation (back-translations) to Norwegian was done by NKVTS. Each measure has 4-items that are scored from 1 (completely disagree) to 5 (completely agree). Average scores are calculated for each measure. The questions will be posed one time to all participating therapists, prior to recruiting first family for SC-TF-CBT.
Intervention Appropriateness Measure (IAM) | Baseline (T0)
  Intervention Appropriateness Measure (IAM) is one of three related instruments (acceptability, appropriateness, and feasibility) developed to fill a need for measures to predicting outcomes, for instance when a treatment is about to be introduced in a new context (Weiner et al., 2017). According to the developers, the measures can be used together or separately. The present research will use the measures, which are scored separately, together to predict how Stepped-Care TF-CBT might suit a Norwegian context. Translation (back-translations) to Norwegian was done by NKVTS. Each measure has 4-items that are scored from 1 (completely disagree) to 5 (completely agree). Average scores are calculated for each measure. The questions will be posed one time to all participating therapists, prior to recruiting first family for SC-TF-CBT.
Feasibility of Intervention Measure (FIM) | Baseline (T0)
  Feasibility of Intervention Measure (FIM) is one of three related instruments (acceptability, appropriateness, and feasibility) developed to fill a need for measures to predicting outcomes, for instance when a treatment is about to be introduced in a new context (Weiner et al., 2017). According to the developers, the measures can be used together or separately. The present research will use the measures, which are scored separately, together to predict how Stepped-Care TF-CBT might suit a Norwegian context. Translation (back-translations) to Norwegian was done by NKVTS. Each measure has 4-items that are scored from 1 (completely disagree) to 5 (completely agree). Average scores are calculated for each measure. The questions will be posed one time to all participating therapists, prior to recruiting first family for SC-TF-CBT.
Child and Adolescent Social Support Scale (CASSS 2000) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The Child and Adolescent Social Support Scale (CASSS 2000) is a scale consisting of four modules. In this study only one of the modules will be included; the children's self-reported experience of social support from the parents. This sub-scale consists of 12 questions. CASSS is a validated instrument for 8-11 year olds (Malecki & Demaray, 2002). The research group has translated the scale in collaboration with the developers, with independent translation back to English (back-translation) to ensure the quality. The 12 items are scored from 1 (never) to 6 (always).
Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) | T1 (day of treatment start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  Children's Post-Traumatic Cognitions Inventory Short (CPTCI-S) measures inappropriate cognitions / thoughts after trauma. The original scale is based on 25 questions, but in this project a 10-item short-version will be used. This is validated for children aged 7-17 years (McKinnon et al., 2016). The 10 items are scored from 1 (don't agree at all) to 4 (agree a lot).
Client Satisfaction Questionnaire (CSQ-8) | T3 (12-15 weeks) or before if treatment ends early.
  The Client Satisfaction Questionnaire (CSQ) has been used to evaluate the parents' satisfaction with Trinnvis TF-CBT in previous studies (Salloum et al., 2014). The 8 items are scored from 4 (excellent) to 1 (poor).
Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) | CGI-S: T0 (baseline), T2 (6-9 weeks), T3 (12-15 weeks). CGI-I: T1 (start-up), P2 (2 weeks), P3 (4 weeks), T2 (6-9 weeks), T3 (12-15), 24-27 weeks (T4). CGI-I from caregiver only collected during 7 telephonecalles inbetween sessions with the therapist.
  Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) consists of one single question each and are used to make a simple assessment of the condition and level of functioning in children at the first meeting and subsequently to assess changes in condition and functioning at later meetings. Both the children and the caregivers will respond, in addition to the therapist (Busner & Targum, 2007). The wording of the questions can easily accommodate different types of patients. CGI has been used in a variety of populations, including children receiving Stepped Care TF-CBT (Salloum et al., 2014), patients with social anxiety (Zaider, Heimberg, Fresco, Schneier, & Liebowitz, 2003) and bipolar disorder (Spearing, Post, Leverich, Brandt, & Nolen, 1997). CGI-S is scored 0 (no symptoms) to 6 (extremely ill). CGI-I is scored from 8 (extreme/serious worsening) to 1 (no symptoms).
Expectancy Rating Form (ERF) | T1 (at treatment start-up)
  ERF originally consists of 5 questions (Borkovec & Nau, 1972). The first 3 questions have previously been used to assess the expectations and trust of Stepped Care TF-CBT prior to initiation of the intervention (Salloum et al., 2014). The questions were adapted from Borkovec and Nau (1972). The project group has made a cross-checked translation of the US version to Norwegian. Items 1-4 are scored from 1 (not at all) to 10 (very). Item 5 is scored on an 11-point scale from 0% to 100% expected improvement.
Multidimensional Scale of Perceived Social Support (MSPSS) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), T4 (24-27 weeks)
  The Multidimensional Scale of Perceived Social Support (MSPSS) consists of 12 questions that reflect experienced support from family, friends and other important people. The scale is validated in several languages (Kazarian & McCabe, 1991; Pedersen, Spinder, Erdman, & Denollet, 2009; Zimet, Dahlem, Zimet, & Farley, 1988; Zimet, Powell, Farley, Werkman, & Berkoff, 1990). The Norwegian translation is done at the University of Bergen and is used in Norwegian context (Steine et al., 2012). The 12 items are scored from 1 (strongly disagree) to 7 (strongly agree).
Parental Emotional Response Questionnaire (PERQ) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The Parental Emotional Response Questionnaire (PERQ) contains 15 questions concerning parents' reactions and feelings in relation to what the child has experienced/ been exposed to, such as guilt, sadness, anger and shame (Mannarino & Cohen, 1996). The scale has shown good validity in studies of parents with children in the age group 7-12 years (Mannarino & Cohen, 1996). PERQ has previously been used in a Norwegian context (Holt, Jensen, & Wentzel-Larsen, 2014). The 15 items are scored from 1 (never) to 5 (always).
Parental Stress Scale (PSS) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The Parental Stress Scale (PSS) consists of 18 questions measuring both the positive aspects of being a parent and experienced stress in parenting (Berry & Jones, 1995). The scale is suitable for use by both guardians and children in clinical trials and in normal selections, and has been used in several countries (Louie, Cromer, & Berry, 2017; Oronoz, Alonso-Arbiol, & Balluerka, 2007) and has also been used in Norway (Nordahl, Zambrana, & Forgatch, 2016). Translation to Norwegian has been done by the National Development Center for Children and Young People (NUBU). The 18 items are scored from 1 (strongly disagree) to 5 (strongly agree).
Pediatric Symptom Checklist (PSC-17) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  Pediatric Symptom Checklist (PSC-17) is a measure of child behavior to be filled out by parents. PSC-17 is a short-form of PSC-34 and contains questions that will measure the attention (such as ability to concentrate), externalizing behavior (such as outward behavior) and internalizing behavior (like anxiety). The PSC-17 has proved to be a good measure compared to longer scales (Gardner, Lucas, Kolko, & Campo, 2007). The scale has been translated into Norwegian by the research group and the Norwegian text has been translated back to English to check the translation (back-translation). The 17 items are scored from 0 (never) to 2 (often).
PTSD Checklist for DSM-5 (PCL-5) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The PTSD Checklist for DSM-5 (PCL-5) consists of 20 questions based on the criteria for PTSD diagnosis in DSM-5 (Weathers, Litz, Herman, Huska, & Keane, 1993). PCL-5 has been translated into Norwegian and validated in Norwegian context (Hem, Hussain, Wentzel-Larsen, & Heir, 2012). The 20 items are scored from 0 (not at all) to 4 (very much).
Short Moods and Feeling Questionnaire (SMFQ) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks)
  The Short Moods and Feeling Questionnaire (SMFQ) consists of 13 questions and is a short version of a longer scale with 54 questions (Moods and Feeling Questionnaire). The questions measure symptoms of depression and are answered by the children. The scale has been validated internationally among children aged 7-11 years (Sharp, Goodyer, & Croudace, 2006), 8-16 years (Angold, Costello, Messer, & Pickles, 1995) and in Norway for the age group 7-17 years (Sachser et al., 2017). The 13 items are scored 0 (not correct) to 2 (correct).
Stressful Life-Events Screening Questionnaire (SLESQ) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The Stressful Life-Events Screening Questionnaire (SLESQ) is a checklist of 15 points that reveals stressful events, such as serious illness, loss of family member in accident, rape and violence (Goodman, Corcoran, Turner, Yuan, & Green, 1998). The checklist has good validity in several cultures (Green, Chung, Daroowalla, Kaltman, & DeBenedictis, 2006) and has been adapted to Norwegian conditions and validated (Thoresen & Øverlien, 2009). The 15 items are answered "yes" or "no."
Symptom Check-list-10 (SCL-10) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The Symptom Check-list-10 (SCL-10) consists of 10 questions that measure anxiety and depression symptoms. SCL-10 is a short version of SCL-90 (Derogatis & Cleary, 1977) and is a widely used and validated scale in Norwegian context (Strand, Dalgard, Tambs, & Rognerud, 2003). The 10 items are scored 1 (a bit bothered) to 4 (not very).
Therapeutic Alliance Scale for Children (TASC): Therapist-Caregiver | P1 (after first session), P2 (2 weeks), P3 (4 weeks), P4/T2 (6-9 weeks)
  The Therapeutic Alliance Scale for Children (TASC) measures how the collaboration is between the therapist and the parent/ guardian (Shirk & Saiz, 1992). It is found in several variants. The scales have been translated and adapted to Norwegian conditions by NKVTS (Ormhaug, Jensen, Wentzel-Larsen, & Shirk, 2014).The 12 items are scored from 1 (not correct at all) to (entirely correct).
Therapeutic Alliance Scale for Children (TASC): Caregiver-Therapist | P1 (after first session), P2 (2 weeks), P3 (4 weeks), P4/T2 (6-9 weeks)
  The Therapeutic Alliance Scale for Children (TASC) measures how the collaboration is between the parent/ caregiver and the therapist (Shirk & Saiz, 1992). There are several variants of the scale. The scales have been translated and adapted to Norwegian conditions by NKVTS (Ormhaug, Jensen, Wentzel-Larsen, & Shirk, 2014). The 14 items are scored 1 (not at all correct) to (entirely correct).
Therapy Satisfaction: 3 questions | T3 (12-15 weeks) or before if treatment ends early.
  Therapy satisfaction is assessed through 3 questions focusing on the therapy experience (liked coming to the therapist, if coming there helped, and the idea of coming again). The three items are scored from 1 (all the time) to 4 (not at all).
Therapeutic Alliance Scale for Children (TASC): Caregiver-Child | P2 (2 weeks), P3 (4 weeks), P4/T2 (6-9 weeks)
  The Therapeutic Alliance Scale for Children (TASC): Caregiver-Child is an adaptation from the original scale developed by (Shirk & Saiz, 1992), and is designed to assess the working alliance with the child as experienced by the caregiver during the home-based exercises. The 7 items are scored from 1 (not correct at all) to (entirely correct).
Therapeutic Alliance Scale for Children (TASC): Child-Caregiver | P2 (2 weeks), P3 (4 weeks), P4/T2 (6-9 weeks)
  The Therapeutic Alliance Scale for Children (TASC): Child-Caregiver is an adaptation from the original scale developed by (Shirk & Saiz, 1992), and is designed to assess the working alliance with the caregiver as experienced by the child during the home-based exercises. The 7 items are scored from 1 (not correct at all) to (entirely correct).
KIDSCREEN School environment module | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The school environment module (6 items) has been included from the KIDSCREEN-52 (Haraldstad et al, 2011), and measures health-related quality of life in relation to the school environment. The response scale has 5 options ranging from not at all to extremely.
Children's somatic symptoms inventory short form (CSSI-8) | T1 (start-up), T2 (6-9 weeks), T3 (12-15 weeks), 24-27 weeks (T4)
  The CSSI-8 (Walker et al, 2016) is derived from the Child Somatization Inventory (CSI-24) and assesses how much the children had been botheres by somatic symptoms. Responses were scored using a four-point Likert scale ranging from 1 (not at all) to 4 (a whole lot).
Barriers for treatment | T1 (start-up)
  A checklist of 9 potential barriers for completing treatment was constructed based on existing measures of barriers, and adapted to the conditions of the study. The list includes illness in the family, work-situation, family stress, economic difficulties and more.
Leadership Implementation Scale (ILS) | Baseline (T0)
  The ILS assesses the degree to which a leader is proactive, knowledgeable, supportive, and perseverant in regard to implementation (Aarons 2014). The scale consists of 12 items and is rated from 0 (Not at all) to 4 (Very great extent).

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Skjærvø, PhD, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (1):
- Norwegian Center for Violence and Traumatic Stress Studies, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salloum A, Scheeringa MS, Cohen JA, Storch EA. Development of Stepped Care Trauma-Focused Cognitive-Behavioral Therapy for Young Children. Cogn Behav Pract. 2014 Feb 1;21(1):97-108. doi: 10.1016/j.cbpra.2013.07.004. PMID 25411544
- [Derived] Ormhaug SM, Skjaervo I, Dyrdal GM, Fagermoen EM, Haabrekke KJ, Jensen TK, Knutsen ML, Naess A, Paivarinne HM, Martinsen M. Stepping Together for Children After Trauma (ST-CT): Feasibility and Predictors of Outcome of a Parent-led, Therapist Assisted Treatment. Res Child Adolesc Psychopathol. 2024 Sep;52(9):1413-1425. doi: 10.1007/s10802-024-01199-5. Epub 2024 May 13. PMID 38739305
- [Derived] Fagermoen EM, Skjaervo I, Birkeland MS, Jensen TK, Ormhaug SM. The bidirectional associations between caregiver and child symptoms in the parent-led treatment stepping together for children after trauma. Behav Res Ther. 2024 Feb;173:104459. doi: 10.1016/j.brat.2023.104459. Epub 2023 Dec 16. PMID 38128401
- [Derived] Fagermoen EM, Skjaervo I, Jensen TK, Ormhaug SM. Parent-led stepped care for traumatised children: parental factors that predict treatment completion and response. Eur J Psychotraumatol. 2023;14(2):2225151. doi: 10.1080/20008066.2023.2225151. PMID 37366166
- [Derived] Fagermoen EM, Jensen TK, Martinsen M, Ormhaug SM. Parent-Led Stepped Care Trauma Treatment: Parents' Experiences With Helping Their Child Recover. J Child Adolesc Trauma. 2023 Mar 31;16(4):1-13. doi: 10.1007/s40653-023-00537-x. Online ahead of print. PMID 37359465